CLINICAL TRIAL: NCT00124202
Title: Effect of a Fatty Meal on Cannulation at Endoscopic Retrograde Cholangiopancreatography
Brief Title: Effect of a Fatty Meal on Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Dr. Qiang Cai MD/PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 229-2003
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Biliary Tract Disease
Keywords: a fatty meal; ERCP
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- a fatty meal vs normal saline (Placebo Comparator): Approximately one hour before ERCP procedure, patient will have a fatty meal in the study group and normal saline in control group
  Interventions: Behavioral: a fatty meal

INTERVENTIONS:
Behavioral: a fatty meal — Approximately one hour before ERCP procedure, patient will have a fatty meal in the study group and normal saline in control group

SUMMARY:
This study is to determine if a fatty meal would improve the ERCP procedure.

DETAILED DESCRIPTION:
A fatty meal is a potent stimulator of cholecystikinin (CCK) in human body. The biological effect of CCK is increasing bile secretion and relaxing the sphincter of Oddi. Theoretically, a fatty meal should facilitate the effect on cannulation at ERCP. If a fatty meal can make the major papilla cannulation easier, it may significantly shorten the procedure time for ERCP and even decrease complications of the procedure, since the complication rate of post-ERCP is positively related to the time of the procedure.

Comparison: Approximately one hour before ERCP procedure, patient will have a fatty meal in the study group and normal saline in control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years and older, who are scheduled for ERCP at Emory University Hospital and signed consent before the procedure.

Exclusion Criteria:

* Patients with a known allergy to milk or those who choose not to sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
a fatty meal in the study group and normal saline in control group | the procedure time for ERCP

SECONDARY OUTCOMES:
follow up within 3 days for complication with relation to the cannulation time | within 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Cai, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine; Emory University Hospital, Atlanta, Georgia, United States